CLINICAL TRIAL: NCT02818751
Title: Neurofunctional Predictors of Escitalopram Treatment Response in Adolescents With Anxiety
Acronym: FiESTAA
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Cincinnati (Other)
Collaborators: National Institute of Mental Health (NIMH) (NIH)
Responsible Party: Principal Investigator, Jeffrey Strawn, MD, Associate Professor of Psychiatry, University of Cincinnati
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: Strawn FiESTAA; K23MH106037 (NIH)
Record Dates: First submitted 2016-06-02; First posted 2016-06-30 (Estimated); Last update posted 2020-11-06 (Actual); Status verified 2020-11

CONDITIONS: Anxiety
Keywords: Anxiety; Adolescents with Anxiety
MeSH Terms: conditions — Anxiety Disorders | interventions — Escitalopram; Sugars

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- Escitalopram (Experimental): Patients being randomized to receive escitalopram, at an initial dose of 5 mg (oral) daily for 2 days. On day 3, escitalopram will be increased to 10 mg daily and continued for 7 days. Then, on day 10, escitalopram will be increased to 15 mg. At the week 4 visit, the dose of escitalopram may be increased to 20 mg, based on the investigator's clinical judgment and if significant anxiety symptoms are still present.
  Interventions: Drug: Escitalopram
- Placebo (Placebo Comparator): Patients will receive placebo (sugar pill) at an initial dose of 5 mg daily for 2 days. On day 3, placebo will be increased to 10 mg daily and continued for 7 days to match the experimental group.
  Interventions: Other: Placebo
- Healthy Controls (No Intervention): Healthy adolescents will receive fMRI scans at the same time points, which will provide assessments of the stability of neurophysiologic measures and will be used to adjust and interpret comparisons within the patients (i.e., whether patient values are changing toward or away from those of healthy adolescents).

INTERVENTIONS:
Drug: Escitalopram — Patients being randomized to receive escitalopram.
  Other Names: Lexapro
  Arms: Escitalopram
Other: Placebo — Patients being randomized to receive placebo.
  Other Names: Sugar Pill
  Arms: Placebo

SUMMARY:
Neurofunctional Predictors of Escitalopram Treatment Response in Adolescents with Anxiety. To determine the effects of escitalopram on functional activation patterns during a Continuous Performance Task with Emotional and Neutral Distracters, the CPT-END. To examine baseline functional activity and functional connectivity profiles in the ventrolateral prefrontal cortex as markers of subsequent treatment response to escitalopram in adolescents with generalized anxiety disorder (GAD). To use proton magnetic resonance spectroscopy (1H MRS) to examine glutamatergic and γ-aminobutyric acid (GABA)-related abnormalities in the anterior cingulate in adolescents with GAD as compared to healthy adolescents.

DETAILED DESCRIPTION:
The long-term goal of this study is to explore the neurobiological basis of generalized anxiety disorder (GAD) using a validated functional MRI (fMRI) paradigm and functional connectivity analyses with a cohort of GAD patients and healthy subjects and generating feasibility and preliminary data regarding treatment-related effects of escitalopram on brain functional activation and Fc patterns in pediatric GAD. An additional goal is to identify biological markers in saliva and urine that will predict treatment response in pediatric subjects with GAD. The central hypothesis of this proposal is that core dysfunction within the prefrontal-amygdala network, which the investigators and others have observed in GAD, will be normalized by successful treatment. The rationale underlying this hypothesis is that, despite the high prevalence of GAD, there is a need to understand its neurobiology and to identify biomarkers of treatment response and the mechanisms by which selective serotonin reuptake inhibitors (SSRIs) putatively effect changes in the neurocircuitry of pediatric GAD.

ELIGIBILITY:
Inclusion Criteria:

Inclusion - Anxiety Subjects:

* Diagnostic and Statistical Manual-IV (Text Revision) criteria for generalized anxiety disorder diagnosed by the Anxiety Disorders Interview Schedule (ADIS-IV)
* Baseline Pediatric Anxiety Rating Scale (PARS) score ≥15 at baseline
* Ages 12-17 years 11 months old
* Fluent in English
* Provision of written informed consent by a legal guardian and written assent by the subject
* Tanner scale stages II-V, in order to include only post-pubescent subjects and minimize brain changes associated with the onset of puberty
* Does not have a history of intolerance, non-response or hypersensitivity to escitalopram
* No co-occurring Diagnostic and Statistical Manual-IV (Text Revision) diagnosis mood (except dysthymia, depression not otherwise specified), eating, pervasive developmental disorder or psychotic disorders
* Subjects will be excluded if there are any lifetime diagnosis of mental retardation (intelligence quotient < 70)
* Subjects with any history of alcohol or drug dependence or any alcohol abuse within the past 6 months (nicotine dependence is permitted) will be excluded
* No new psychotherapy will be permitted during study participation and if the patient is engaged in psychotherapy, it must have been stable for 1 month prior to baseline
* Females will not be eligible to participate if pregnant, breast feeding or lactating.

Inclusion - Healthy Subjects:

* Ages of 12-17 years and 11 months
* No history of any Diagnostic and Statistical Manual-IV (Text Revision) Axis I disorders (nicotine dependence is permitted)
* No first-degree relatives with an affective or psychotic disorder
* No medications with central nervous system effects within 5 half-lives
* Fluent in English
* Tanner stage II-V
* Provision of informed consent and assent.

Exclusion Criteria:

Exclusion - Generalized Anxiety Disorder Patients & Healthy Subjects:

* Contraindication to an magnetic resonance imaging (MRI) scan (e.g., braces or claustrophobia)
* An unstable medical or neurological illness that could influence fMRI or magnetic resonance spectroscopy results
* Subjects will be excluded if there are any lifetime diagnosis of mental retardation or intelligence quotient < 70)
* A positive pregnancy test
* Adolescents will be excluded for treatment with a medication with central nervous system effects that requires more than 5 days of a screening period in order to minimize the length of time between screening and baseline and maximize patient safety, while recognizing that a longer taper period is required of some medications
* Adolescents with any history of major medical or neurological disorders that may result in neurofunctional or neurochemical abnormalities including loss of consciousness for >10 minutes will be excluded
* No co-occurring Diagnostic and Statistical Manual-IV (Text Revision) diagnosis mood (other than dysthymia or Depression Not Otherwise Specified), eating, pervasive developmental disorder or psychotic disorders
* Subjects will be excluded if there are any lifetime diagnosis of mental retardation or intelligence quotient < 70
* Subjects with any history of alcohol or drug dependence or any alcohol abuse within the past 6 months (nicotine dependence is permitted) will be excluded
* No new psychotherapy will be permitted during study participation and if the patient is engaged in psychotherapy, it must have been stable for 1 month prior to baseline
* Females will not be eligible to participate if pregnant, breast feeding or lactating
* The patient lives >100 miles from the University of Cincinnati or is not able to attend follow-up visits

Ages: 12 Years to 17 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 84 (Actual)
Dates: Start 2015-05 (Actual); Primary Completion 2019-05 (Actual); Study Completion 2020-05 (Actual)

PRIMARY OUTCOMES:
Early escitalopram-related functional brain activity changes during emotional processing | From baseline to week 2 of treatment
  To determine if escitalopram treatment (over a 2 week period) increases functional brain activation during the processing of emotional images while performing a continuous processing task with emotional and neutral distracters (CPT-END) (also over a 2 week period).

SECONDARY OUTCOMES:
Change in functional activity in the ventrolateral prefrontal cortex (from baseline to week 2) and improvement in Pediatric Anxiety Rating Scale score (at week 8/early termination) | from baseline to week 8 (or early termination)
  To determine if the change in functional activity in the ventrolateral prefrontal cortex (from baseline to week 2) predicts improvement in Pediatric Anxiety Rating Scale score from baseline to week 8/early termination.
Change in functional connectivity between the ventrolateral prefrontal cortex and the amygdala (from baseline to week 2) and improvement in Pediatric Anxiety Rating Scale score (at week 8/early termination) | from baseline to week 8 (or early termination)
  To determine if the change in functional connectivity between the ventrolateral prefrontal cortex and the amygdala (from baseline to week 2) predicts improvement in Pediatric Anxiety Rating Scale score from baseline to week 8/early termination.
Change in glutamate concentrations in the anterior cingulate cortex predict improvement in Pediatric Anxiety Rating Scale score from baseline to week 8/early termination. | from baseline to week 8 (or early termination)
  To determine if change in glutamate concentrations in the anterior cingulate cortex predict improvement in Pediatric Anxiety Rating Scale score from baseline to week 8/early termination.
Change in γ-aminobutyric acid concentrations in the anterior cingulate (from baseline to week 2) predicts improvement in Pediatric Anxiety Rating Scale score from baseline to week 8 (or early termination) | from baseline to week 8 (or early termination)
  To determine if the change in γ-aminobutyric acid concentrations in the anterior cingulate (from baseline to week 2) predicts improvement in Pediatric Anxiety Rating Scale score from baseline to week 8 (or early termination)

CONTACTS AND LOCATIONS:
Overall Officials: Jeffrey Strawn, Principal Investigator — University of Cincinnati
Locations (1):
- University of Cincinnati, Department of Psychiatry & Behavioral Neuroscience, Cincinnati, Ohio, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Strawn JR, Mills JA, Schroeder H, Mossman SA, Varney ST, Ramsey LB, Poweleit EA, Desta Z, Cecil K, DelBello MP. Escitalopram in Adolescents With Generalized Anxiety Disorder: A Double-Blind, Randomized, Placebo-Controlled Study. J Clin Psychiatry. 2020 Aug 25;81(5):20m13396. doi: 10.4088/JCP.20m13396. PMID 32857933
- [Result] Lu L, Li H, Mills JA, Schroeder H, Mossman SA, Varney ST, Cecil KM, Huang X, Gong Q, Levine A, DelBello MP, Sweeny JA, Strawn JR. Greater Dynamic and Lower Static Functional Brain Connectivity Prospectively Predict Placebo Response in Pediatric Generalized Anxiety Disorder. J Child Adolesc Psychopharmacol. 2020 Dec;30(10):606-616. doi: 10.1089/cap.2020.0024. Epub 2020 Jul 24. PMID 32721213
- [Derived] Marusak HA, Zundel CG, Shakir T, Ely SL, Carpenter C, Shampine M, Tamimi R, Matsko M, Rogers S, Losiowski J, O'Mara E, Jaster AM, Sharma K, deRoon-Cassini TA, Hillard CJ, Schroeder HK, Mills JA, Strawn JR, Barcelona J. Circulating endocannabinoids in children and adolescents: associations with anxiety and the impact of selective serotonin reuptake inhibitors. Neuropsychopharmacology. 2025 Sep;50(10):1606-1614. doi: 10.1038/s41386-025-02155-7. Epub 2025 Jun 27. PMID 40579470
- [Derived] Lu L, Li H, Baumel WT, Mills JA, Cecil KM, Schroeder HK, Mossman SA, Huang X, Gong Q, Sweeney JA, Strawn JR. Acute neurofunctional effects of escitalopram during emotional processing in pediatric anxiety: a double-blind, placebo-controlled trial. Neuropsychopharmacology. 2022 Apr;47(5):1081-1087. doi: 10.1038/s41386-021-01186-0. Epub 2021 Sep 27. PMID 34580419
- [Derived] Lu L, Mills JA, Li H, Schroeder HK, Mossman SA, Varney ST, Cecil KM, Huang X, Gong Q, Ramsey LB, DelBello MP, Sweeney JA, Strawn JR. Acute Neurofunctional Effects of Escitalopram in Pediatric Anxiety: A Double-Blind, Placebo-Controlled Trial. J Am Acad Child Adolesc Psychiatry. 2021 Oct;60(10):1309-1318. doi: 10.1016/j.jaac.2020.11.023. Epub 2021 Feb 4. PMID 33548492